CLINICAL TRIAL: NCT01126515
Title: MRI & CT Angiogram and Hyperbaric Oxygen in Chronic Stable Brain Injury
Brief Title: Functional and Anatomical Magnetic Resonance Imaging (MRI) of Chronic Brain Injury and Hyperbaric Oxygen (HBO2) Study Subjects
Acronym: HYBOBI-MRI
Status: Completed | Type: Observational
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: Deseret Foundation (Other)
Responsible Party: Principal Investigator, Lindell Weaver, Medical Director, Hyperbaric Medicine, Intermountain Health Care, Inc.
Other Study IDs: 1004120
Record Dates: First submitted 2010-03-01; First posted 2010-05-19 (Estimated); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Brain Injury; Sequelae; Stroke; Anoxia; Trauma
Keywords: brain injury; sequelae; stroke; anoxia; trauma
MeSH Terms: conditions — Brain Injuries; Stroke; Hypoxia; Wounds and Injuries | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hyperbaric oxygen: In this open-label feasibility study, all subjects will receive 60 hyperbaric oxygen sessions (100% oxygen, 1.5 atmospheres absolute (atm abs), for 60 minutes), delivered daily, five days per week.
  Interventions: Procedure: Magnetic Resonance Imaging; Procedure: Computed Tomography Angiography

INTERVENTIONS:
Procedure: Magnetic Resonance Imaging — Imaging of the brain without gadolinium will be performed with a 3 Tesla magnetic resonance (MR) System (Intera Achieva 3T; Philips Medical Systems). The protocol will include anatomical sequences, a diffusion tensor imaging sequence with fiber tracking, and auditory, visual, and motor functional magnetic resonance imaging (MRI).
  Other Names: MRI; fMRI
Procedure: Computed Tomography Angiography — Computed tomography angiography (CTA) with intravenous (IV) contrast will be performed on a 320 head computed tomography (CT) scanner, assessing brain perfusion.
  Other Names: CT; CTA

SUMMARY:
The purpose of this study is to evaluate Brain MRI (Magnetic Resonance Imaging), and Brain CT (Computed Tomography) Angiogram data in subjects who participate in the "Hyperbaric Oxygen for Chronic Stable Brain Injury" (HYBOBI) study. Including information from MRI and CT studies provide information about whether hyperbaric oxygen improves brain function in subjects who have had a brain injury. Subjects will complete MR and CT scans twice during the study. The first MR and CT will be performed prior to the first hyperbaric session of the HYBOBI study, and the second will be performed within two weeks following the last hyperbaric session.

DETAILED DESCRIPTION:
In an ongoing feasibility study (HYBOBI), brain-injured subjects are exposed to hyperbaric oxygen at 1.5 atmospheres for 60 minutes. They receive this exposure five days per week, and receive 60 total sessions. Prior to hyperbaric oxygen, these study subjects have neurologic, cognitive, and functional measures. The measures are repeated at the conclusion of 60 hyperbaric oxygen sessions, and again six months later. The goal of the HYBOBI feasibility study is to learn about these patients and determine possible hyperbaric oxygen effects, if any, to prepare for a blinded randomized controlled clinical trial.

This study adds an imaging component to the HYBOBI study, further investigating brain changes in participants. Participants will undergo Brain MRI (Magnetic Resonance Imaging) using a 3 tesla magnet, and Brain CT (Computed Tomography) Angiogram. Subjects will undergo imaging before receiving hyperbaric oxygen and within 2 weeks of completion of the 60 hyperbaric sessions.

ELIGIBILITY:
Inclusion Criteria:

* Subject has had a brain injury > 12 months
* Subject is >18 years old
* Etiology of brain injury:

  * stroke
  * carbon monoxide
  * anoxia
  * trauma
* Must be able to equalize ears, or have tympanostomy tubes
* Willingness to complete outcome measures and comply with the research protocols
* Commitment to pay the hospital for hyperbaric oxygen
* Subject is enrolled in Hyperbaric Oxygen and Chronic Stable Brain Injury study-clinical trials government ID# NCT00830453.

Exclusion Criteria:

* Glasgow Coma Score <13 at the time of consent
* Poorly controlled seizures
* Inability to participate in outcome assessments (eg: blindness, quadraplegia); Claustrophobia
* Inability to equalize ears
* Inability to protect airway, or requiring frequent suctioning
* Tracheostomy
* Women of child-bearing potential or currently pregnant
* Severe psychiatric disorders
* Taking lithium
* Degenerative mental disease
* Chronic debilitating disease
* Heart failure with ejection fraction <50% or inability to lay supine
* Active malignancy, or prior treatment with cisplatin or bleomycin
* Current recreational drug use
* Consumption of more than the equivalent of 12 beers/week habitually
* Prior treatment with hyperbaric oxygen for chronic brain injury within the last year
* Implanted device that is a contra-indication to MRI
* Inability to travel to Las Vegas, either by car or by air
* Serum creatinine greater than the Intermountain Central Lab normal limit
* Unwillingness or inability to have intravenous contrast.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with chronic brain injury who are enrolled in the HYBOBI study.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2007-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Auditory functional magnetic resonance imaging (fMRI) activation | Within 2 weeks of final hyperbaric session
  The first prime outcome measure will be auditory functional magnetic resonance imaging (fMRI) activation, comparing post-hyperbaric oxygen to pre-hyperbaric oxygen. This is a categorical variable: absent, mild, moderate, normal, and increasing. We will look at the difference between pre-hyperbaric (pre-HBO2) and post-hyperbaric (post-HBO2) scans graphically and descriptively, with the percentage of patients who show any improvement (any change towards normal).
Computed tomography angiography (CTA) Brain Perfusion | Within 2 weeks of the final hyperbaric session
  Pre-hyperbaric (pre-HBO2) computed tomography angiography (CTA) results will be determined to be normal or abnormal, and then compared to the post-hyperbaric (post-HBO2) scan, which will be scored as better, worse, or no change.

SECONDARY OUTCOMES:
MRI Results | Within 2 weeks of the final hyperbaric session
  1. Cortical activation (amount and location) for motor, visual, and olfactory fMRI.
  2. Diffusion tensor imaging (fractional anisotropy differences, number of fiber tracts) within the Corpus Callosum

CONTACTS AND LOCATIONS:
Overall Officials: Susan K Churchill, APRN-NP, Principal Investigator — Intermountain Health Care, Inc.; Lindell K Weaver, MD, Principal Investigator — Intermountain Health Care, Inc.
Locations (1):
- LDS Hospital, Salt Lake City, Utah, United States